CLINICAL TRIAL: NCT06759610
Title: Effect of Tetracycline Socked Pack on Acceleration of Healing During Marsupialization as a Primary Treatment for Locally Invasive Lesion: Single Blinded Randomized Clinical Trial
Brief Title: Effect of Tetracycline Socked Pack on Acceleration of Healing During Marsupialization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Tarek Abdelbarry, Lecturer of Oral and Maxillofacial Surgery, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tetracycline Socked Pack
Record Dates: First submitted 2024-12-28; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-02

CONDITIONS: Ameloblastoma
MeSH Terms: conditions — Ameloblastoma | interventions — Tetracycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): About 7 patients who will be subjected to marsupialization procedure with a tetracycline socked pack during marsupialization
  Interventions: Drug: Tetracyclin
- Group B (Active Comparator): About 7 patients who will undergo conventional marsupialization procedure
  Interventions: Drug: Tetracyclin

INTERVENTIONS:
Drug: Tetracyclin — to evaluate the effect of tetracycline socked pack on acceleration of healing during marsupialization as a primary treatment for locally invasive lesions.
  Other Names: marsupialization procedure

SUMMARY:
Ameloblastoma is an epithelial odontogenic tumor. Although ameloblastoma is classified as a benign tumor, it is locally invasive with high recurrence rate. It accounts for up to 18 % of all oral and odontogenic tumors.

Tetracyclines discovered in 1940s show activity against a wide variety of microorganisms including both Gram-positive and Gram-negative bacteria. Chlamydia, rickettsia, mycoplasmas, and protozoan parasites are also under its spectrum. Mechanism of action of tetracyclines is that it inhibits protein synthesis in bacteria by preventing the association of aminoacyl-tRNA with bacterial ribosome.

DETAILED DESCRIPTION:
Ameloblastoma can be described as a silent lesion, as it grows slowly and usually becomes symptomatic when it reaches a large size. Unicystic ameloblastoma (UA) accounts for about 5 % to 15 % of all ameloblastoma, with reported recurrence rates 10 % to 25%. More than 90 % of unicystic ameloblastoma involve the mandible, mostly the posterior region.

Unicystic ameloblastoma (UA) refers to those lesions that show clinical and radiographic features of an odontogenic cyst but on histological examination show an ameloblastic proliferation into the cystic lumen, confined to the cyst lining, or invade the cystic wall, hence their name are intraluminar, luminar, or mural unicystic ameloblastoma (UA), respectively.

As UA less aggressive and has low recurrence rate than conventional type, conservative approaches have been widely used for treatment of UA such as marsupialization, marsupialization followed by enucleation, or enucleation alone or with adjunctive modalities as bone curettage, or application of liquid nitrogen or carnoy's solution.

Despite progress in reconstructive surgery, extensive jaw resection influences quality of life and causes numerous complications. For this cause particularly, conservative treatment of unicystic ameloblastoma in young patients should be superior choice over other treatment methods. Marsupialization by simple definition, is the creation of a pouch surgically, by removing part of the overlying mucoperiosteoum and accompanying cyst wall; followed by suturing of the incised mucosa with the border of the remaining cyst wall that has been leaved.The reduced tension gives rise to healing and formation of bone with the surrounding bone.

Matrix metalloproteinases (MMPs) are a group of Zn-dependent enzymes which regulate inflammation. Pathologically, the elevation of MMPs causes connective tissue and bone loss in various inflammatory diseases. Tetracyclines are effective inhibitors of mammalian MMPs. Tetracyclines can inhibit both intracellular and extracellular MMPs. Tetracycline inhibits MMPs on specific sites that have been identified as the calcium and zinc-binding site at C-11 and 12.

The anti-inflammatory nature of tetracycline is utilized in the various dermatological diseases and in periodontitis too. The anti-inflammatory property of tetracyclines can be useful in the reduction of postoperative sequalae following extraction.

ELIGIBILITY:
Inclusion Criteria:

* patients (class I category according to American society of anesthesiologists) over 20 years and under 40 years of age, of either gender who are seeking treatment of a painful intra-body mandibular swelling cystic lesions 3 x 4 cm in size with biopsy conformation that the lesion is a Uni-cystic ameloblastoma

Exclusion Criteria:

* any systemic disease that interferes with bone healing,
* patients with significant medical condition,
* alcoholic individuals,
* patients on drugs that affect the central nervous systems,
* patients who reported pregnancy, lactation.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Radiographic assessment CBCT | From baseline to 3 and 6 months after the operation day
  Radiographic assessment evaluate healing process CBCT (Planmeca Promax 3DMid machine, Helsinki Finland) scan will be obtained immediately post-operative ,3 and 6 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: TAREK ABDELBARY, Lecturer, Principal Investigator — Faculty of Dentistry, Minia University
Locations (1):
- Faculty of Dentistry, Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided